CLINICAL TRIAL: NCT01105663
Title: Pharmacologic Impact on Sedation Assessment
Brief Title: Pharmacologic Impact on Sedation Assessments
Acronym: PISA
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-007453; R01HL098087-01 (NIH)
Record Dates: First submitted 2010-03-31; First posted 2010-04-16 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Pediatric Acute Lung Injury
Keywords: sedated; intubated; mechanically ventilated; pediatric; lung injury
MeSH Terms: conditions — Lung Injury | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The primary evaluation will be the assessment of morphine/midazolam pharmacokinetics (PK) and pharmacodynamics (PD). Data from all fully evaluable subjects will be included in the analysis. Analyses will be model based.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sedated, Intubated, Morphine: Subjects will receive morphine/midazolam as part of clinical care. Pharmacokinetic and pharmacogenetic sampling and pharmacodynamic monitoring will occur as indicated. Pharmacokinetic samples will be assayed in the laboratory of the Division of Clinical Pharmacology and Therapeutics. Pharmacogenetic samples will be assayed in the laboratory of the Center for Applied Genomics at CHOP.
  Interventions: Other: Pharmacokinetic Sampling and pharmacogenetic analysis
- Sedated, Intubated, Midazolam: Subjects will receive morphine/midazolam as part of clinical care. Pharmacokinetic and pharmacogenetic sampling and pharmacodynamic monitoring will occur as indicated. Pharmacokinetic samples will be assayed in the laboratory of the Division of Clinical Pharmacology and Therapeutics. Pharmacogenetic samples will be assayed in the laboratory of the Center for Applied Genomics at CHOP.
  Interventions: Other: Pharmacokinetic Sampling and pharmacogenetic analysis

INTERVENTIONS:
Other: Pharmacokinetic Sampling and pharmacogenetic analysis — Pharmacogenetic and pharmacokinetic samples will be obtained from a peripheral catheter, central catheter, or venipuncture coordinated with scheduled phlebotomies. Pharmacokinetic and pharmacogenetic analyses will be performed. Pharmacodynamic data will be collected.
  Other Names: Pharmacokinetic Sampling; pharmacogenetic Sampling

SUMMARY:
PISA is an ancillary study to the NIH funded clinical RESTORE Trial (U01 HL086622). This study will provide data that may allow for improved dosing recommendations in this critically ill population of children.

DETAILED DESCRIPTION:
PISA is an ancillary study to the NIH funded clinical RESTORE Trial (U01 HL086622). This project will use sophisticated modeling and simulation techniques to evaluate the impact of genetics and other variables such as degree of illness, age, weight and organ dysfunction on the pharmacokinetics and pharmacodynamics of morphine and midazolam in children who are mechanically ventilated for respiratory failure, and require sedation. This proposed work will allow the design of a pharmacologic model that can be used to individualize therapy in children requiring mechanical ventilation with the goal of optimizing sedation while minimizing the duration of mechanical ventilation. This study will provide data that may allow for improved dosing recommendations in this critically ill population of children.

ELIGIBILITY:
Inclusion Criteria:• Enrolled in RESTORE clinical trial

* Be greater than or equal to 7 kg
* Receiving morphine and/or midazolam continuous infusions
* Give Informed Consent/Assent

Exclusion Criteria:

* Intubated and mechanically ventilated for immediate post-operative care and stabilization
* Cyanotic heart disease with unrepaired or palliated right to left intracardiac shunt
* History of single ventricle at any stage of repair
* Congenital diaphragmatic hernia or paralysis
* Primary pulmonary hypertension
* Critical airway (e.g., post laryngotracheal construction) or anatomical obstruction of the lower airway (e.g., mediastinal mass)
* Ventilator dependent (including noninvasive) on Pediatric Intensive Care Unit (PICU) admission (chronic assisted ventilation)
* Neuromuscular respiratory failure
* Spinal cord injury above the lumbar region
* Pain managed by patient controlled analgesia (PCA) or epidural catheter
* Family/medical team has decided not to provide full support (patient treatment considered futile)
* Enrolled in any other sedation clinical trial concurrently or within the last 30 days
* Known allergy to any of the study medications.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects must be enrolled in the parent study RESTORE, be at least 10kg, and be receiving either morphine and/or midazolam continuous infusions.
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
In children who are mechanically ventilated, to quantitatively define the heritable factors that underlie the variability in 1) midazolam and 2) morphine exposure and response. | 36-48 months
  This is a pharmacokinetic, pharmacogenetic and pharmacodynamic study examining heritable (specific polymorphisms) on drug exposure, metabolite formation and pharmacodynamic response.

SECONDARY OUTCOMES:
In children who are mechanically ventilated, to quantitatively define the non-heritable factors that underlie the variability in 1) midazolam and 2) morphine exposure and response. | 36-48 months
  Polymorphisms in drug metabolizing systems.

CONTACTS AND LOCATIONS:
Overall Officials: Athena Zuppa, MD MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States